CLINICAL TRIAL: NCT00206180
Title: A Multicenter, Double-Blind, Randomized Trial of the Relationship of Intragastric Acid Control and Healing Status of Moderate and Severe Erosive Esophagitis After Treatment With Esomeprazole Magnesium (NEXIUM®) 10 mg and 40 mg Once Daily
Brief Title: NEXIUM® in the Treatment of Moderate and Severe Erosive Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D9612L00062
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Erosive Esophagitis; Reflux Esophagitis; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux | interventions — Esomeprazole; Dosage Forms

INTERVENTIONS:
Drug: esomeprazole magnesium (oral medication)

SUMMARY:
The purpose of this study is to decide if controlling stomach acid is related to healing of erosive esophagitis after treatment with esomeprazole magnesium (NEXIUM®) 10 mg and 40 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients between the ages of 18 and 75 years
* Patients must have moderate to severe erosive esophagitis

Exclusion Criteria:

* Significant gastrointestinal bleeding
* Severe heart, lung, liver or kidney disease
* Esophagitis not related to acid reflux

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To determine the relationship between 24-hour intragastric pH at Day 5 and healing status of moderate to severe erosive esophagitis, after 4 weeks of treatment with 2 doses of esomeprazole magnesium.

SECONDARY OUTCOMES:
Secondary outcomes and the relationship to pH will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Nexium Medical Science Director, MD, Study Director — AstraZeneca
Locations (39):
- United States (39):
  - Research Site, Alabaster, Alabama
  - Research Site, Anaheim, California
  - Research Site, Dinuba, California
  - Research Site, Fresno, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Bridgeport, Connecticut
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Rome, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Oakbrook Terrace, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Egg Harbor, New Jersey
  - Research Site, Passaic, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, North Providence, Rhode Island
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Ogden, Utah
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Katz PO, Ginsberg GG, Hoyle PE, Sostek MB, Monyak JT, Silberg DG. Relationship between intragastric acid control and healing status in the treatment of moderate to severe erosive oesophagitis. Aliment Pharmacol Ther. 2007 Mar 1;25(5):617-28. doi: 10.1111/j.1365-2036.2006.03235.x. PMID 17305763